CLINICAL TRIAL: NCT05054166
Title: Efficacy of Everolimus-containing Chemotherapy in HER2 Negative Metastatic Breast Cancer Patients With PI3K/AKT/mTOR Mutations: A Retrospective Study
Brief Title: Efficacy of Everolimus-containing Chemotherapy in HER2- mBC Patients With PI3K/AKT/mTOR Mutations Study
Status: Completed | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wen-Ming Cao, Professor, Zhejiang Cancer Hospital
Other Study IDs: EVE-CWM-01
Record Dates: First submitted 2021-09-02; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer; PI3K/AKT/mTOR Pathway Mutation; Everolimus
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

INTERVENTIONS:
Other: No intervention, it was a retrospective study. — This study aimed to retrospectively investigate the efficacy of the everolimus-containing chemotherapy in metastatic breast cancer patients with PI3K/AKT/mTOR mutations.There was no intervention.

SUMMARY:
The study aimed to investigate the efficacy of the everolimus-containing chemotherapy in metastatic breast cancer patients with PI3K/AKT/mTOR mutations.14 cases of HER2- metastatic breast cancer patients with PI3K/AKT/mTOR mutations treated with everolimus-containing chemotherapy were retrospectively analyzed.The genetic profile in PI3K/AKT/mTOR pathway was studied.

DETAILED DESCRIPTION:
The PI3K/AKT/mTOR pathway is frequently altered in breast cancer. Everolimus is a selective inhibitor of mammalian target of Rapamycin (mTOR).The benefit of everolimus in metastatic breast cancer patients with PI3K/AKT/mTOR mutations remains unclear, especially in TNBC patients. The study aimed to investigate the efficacy of the everolimus-containing chemotherapy in metastatic breast cancer patients with PI3K/AKT/mTOR mutations.

14 cases of HER2- metastatic breast cancer participants with PI3K/AKT/mTOR mutations treated with everolimus-containing chemotherapy were retrospectively analyzed.The genetic profile in PI3K/AKT/mTOR pathway was studied.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HER2- metastatic breast cancer
2. Patients with PI3K/AKT/mTOR mutation

Exclusion Criteria:

1. Patients treated with endocrinotherapy and everolimus.
2. The efficacy evaluation could not be available.

Ages: 29 Years to 66 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2- metastatic breast cancer patients with PI3K/AKT/mTOR mutations treated with everolimus-containing chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
PFS | The PFS was defined as the interval from the date of taking the everolimus-containing chemotherapy to the date of the first occurrence of disease progression or death from any cause,whichever came first, assessed up to 24 months.
  Progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-jia Wang, Dr, Study Director — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China